CLINICAL TRIAL: NCT03103230
Title: Recherche de Marqueurs Pronostiques électro-physiologiques précoces Chez l'Aphasique après un Accident Vasculaire cérébral.APHA-TMS
Brief Title: Electro-physiological Signs to Prognostic Aphasia Recovery After a Stroke
Acronym: APHA-TMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX2013/08
Record Dates: First submitted 2015-01-15; First posted 2017-04-06 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2017-03

CONDITIONS: Stroke; Aphasia
Keywords: Motor evoked potentials; aphasia; prognosis; stroke
MeSH Terms: conditions — Stroke; Aphasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Motor Evoked Potentials (Experimental): Patients with aphasia after a stroke
  Interventions: Device: Cortical magnetic stimulation

INTERVENTIONS:
Device: Cortical magnetic stimulation — Motor Evoked Potentials of lips and hand recorded after cortical magnetic stimulation

SUMMARY:
The purpose of this study is to study, among the aphasic person, if motor function ( studied by Motor Evoked Potentials) performed within the first 14 days after a stroke can predict a good recovery from aphasia 6 months of the initial episode.

DETAILED DESCRIPTION:
• Background : Stroke affects approximately 130,000 people per year and communication disorders occur in 35% of cases, resulting in left brain damages. Aphasia is the main cause of these disorders. It is a sign of poor prognosis in the functional recovery after stroke. Recent studies have attempted to establish early clinical prognostic criteria to establish a predictive model of aphasia recovery. The issue of the possibility of prediction is important and can influence the rehabilitation treatment decided in the early days after stroke, with adequate guidance in rehabilitation structures.

There are close links between motor system and language, either at production or comprehension, and more particularly concerning the motricity of the hand or lips. The cortical excitability of motor areas of the right upper limb is thus modified by the language in healthy subjects, but also in the aphasic person.

* Purpose : The main: to study, among the aphasic person, if Motor Evoked Potentials (MEP) performed within the first 14 days after a stroke can predict a good recovery from aphasia 6 months of the initial episode.
* Detailed description: All aphasic stroke patients with ischemic or hemorrhagic damages will be proposed for inclusion. All patients will benefit in the acute phase of an aphasia evaluation, and a clinical evaluation. All patients will have a study of motor evoked potentials (abductor pollicis brevis and orbicularis oris) less than 14 days from stroke. The investigators will evaluate the aphasia 3 and 6 months after stroke, to determinate if MEP can predict a good recovery of aphasia.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a left stroke (first clinical episode deficit) imaging confirmed.
* With aphasia (-1 language analysis in the acute phase and severity of the questionnaire LAST (Flamand-Roze, Falissard et al. 2011))
* Right-handed (Edinburgh Handedness Inventory)
* Free of dementia before stroke
* Older than 18 years
* French
* Able to hold a sitting in chair.
* Included in maximum 14 days after stroke
* Patient social security system
* Free Consent, informed writing signed by the participant or the person of confidence and the investigator (no later than the day of inclusion and before any examination required by research)

Exclusion Criteria:

* Refusal of the consent
* Impaired alertness
* Dementia prior to stroke
* Illiteracy
* Severe dysarthria
* Previous psychiatric history requiring hospitalization in a specialized environment for more than two months
* Pregnant
* Major visual or auditory perceptual disorder
* Previous epilepsy or seizures in hyperacute phase of stroke
* Treatment strongly interacting with GABAergic or glutamatergic system
* Contraindication to MEP: clip intracranial ferromagnetic pacemakers, cochlear implant, intracerebral stimulator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Evolution of aphasia | 6 months after stroke
  Aphasia Severity Rating Scale (ASRS)

SECONDARY OUTCOMES:
Evolution of aphasia | 3 months after stroke
  Aphasia Severity Rating Scale Score (ASRS)
Pattern of aphasia | 3 & 6 months after stroke
  Boston Diagnostic Aphasia Examination (BDAE) ;
Pattern of aphasia | 3 & 6 months after stroke
  Language Screening Test (LAST b)

CONTACTS AND LOCATIONS:
Overall Officials: GLIZE Bertrand, MD, Principal Investigator — University Hospital Bordeaux, France, EA 4136 Univ. Bordeaux, France; PICAT Quitterie, MD, Study Chair — Unité de Soutien Méthodologique à la Recherche Clinique
Locations (1):
- CHU de Bordeaux, Bordeaux, France

REFERENCES:
- [Result] Dickey, L., A. Kagan, et al. (2010).
- [Result] El Hachioui, H., H. F. Lingsma, et al. (2013).
- [Result] Fadiga L, Craighero L, Buccino G, Rizzolatti G. Speech listening specifically modulates the excitability of tongue muscles: a TMS study. Eur J Neurosci. 2002 Jan;15(2):399-402. doi: 10.1046/j.0953-816x.2001.01874.x. PMID 11849307
- [Result] Meister IG, Wilson SM, Deblieck C, Wu AD, Iacoboni M. The essential role of premotor cortex in speech perception. Curr Biol. 2007 Oct 9;17(19):1692-6. doi: 10.1016/j.cub.2007.08.064. Epub 2007 Sep 27. PMID 17900904
- [Result] Meister IG, Sparing R, Foltys H, Gebert D, Huber W, Topper R, Boroojerdi B. Functional connectivity between cortical hand motor and language areas during recovery from aphasia. J Neurol Sci. 2006 Sep 25;247(2):165-8. doi: 10.1016/j.jns.2006.04.003. Epub 2006 Jun 5. PMID 16737714
- [Result] Meister IG, Buelte D, Staedtgen M, Boroojerdi B, Sparing R. The dorsal premotor cortex orchestrates concurrent speech and fingertapping movements. Eur J Neurosci. 2009 May;29(10):2074-82. doi: 10.1111/j.1460-9568.2009.06729.x. Epub 2009 May 9. PMID 19453637
- [Result] Tokimura H, Tokimura Y, Oliviero A, Asakura T, Rothwell JC. Speech-induced changes in corticospinal excitability. Ann Neurol. 1996 Oct;40(4):628-34. doi: 10.1002/ana.410400413. PMID 8871583